CLINICAL TRIAL: NCT03643770
Title: Effect of a Novel Intervention Using Daily Intermittent Hypoxia and High Intensity Training on Upper Limb Function in Individuals With Spinal Cord Injury
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Zev Rymer, Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: STU 00206035; CDMRP-SC160072 (Other Grant/Funding Number: CDMRP-eBRAP Log Number)
Record Dates: First submitted 2018-03-12; First posted 2018-08-23 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries
Keywords: hypoxia
MeSH Terms: conditions — Spinal Cord Injuries; Hypoxia

STUDY DESIGN:
Intervention Model Description: 4 randomized groups: Acute Intermittent Hypoxia (AIH) treatment, AIH in combination with upper extremity training, Sham AIH therapy in combination with upper extremity training and Sham AIH therapy
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Acute Intermittent Hypoxia (AIH) treatment (No Intervention): The mask will first provide a normoxic air (room air) mixture (FiO2 = 0.21) via the mask. The mask is designed to couple with a universal mask circuit connecting to the air mixture system. The purpose of the mask will be to minimize room air entrainment.
- AIH in combination with upper extremity training (Active Comparator): The mask will first provide a normoxic air (room air) mixture (FiO2 = 0.21) via the mask. The mask is designed to couple with a universal mask circuit connecting to the air mixture system. The purpose of the mask will be to minimize room air entrainment. In addition to this upper extremity training will be given using an upper-limb robotic rehabilitation device.
  Interventions: Combination Product: Upper extremity training/Armeo Spring
- Sham AIH therapy in combination with upper extremity training (Active Comparator): Sham hypoxia followed by upper extremity training will be given using an upper-limb robotic rehabilitation device (Armeo Spring®, Hocoma AG, Switzerland). Armeo Spring is a gravity support system based on an ergonomic arm exoskeleton with integrated springs.
  Interventions: Combination Product: Upper extremity training/Armeo Spring
- Sham AIH therapy (No Intervention): Sham hypoxia

INTERVENTIONS:
Combination Product: Upper extremity training/Armeo Spring — Armeo Spring is a gravity support system based on an ergonomic arm exoskeleton with integrated springs.
  Arms: AIH in combination with upper extremity training; Sham AIH therapy in combination with upper extremity training

SUMMARY:
Currently, there are a variety of approaches utilized in attempts to improve upper extremity function, including: traditional therapy, neuroprostheses, botulinum toxin injections, or surgical interventions. In addition, regenerative and restorative therapies, such as: epidural stimulation, functional electrical stimulation, and stem cell therapies, show promise in animal models, but are not ready for clinical translation. Subsequently, there is a clear need to develop new strategies that can stimulate spinal plasticity and strengthen existing synaptic connections in order to maximize the benefits of training paradigms.

This study proposes the examine the effects of Acute Intermittent Hypoxia (AIH) in combination with upper extremity training, over the course of a month, to evaluate changes in upper extremity function, dexterity, and ability to complete activities of daily living. The use of acute intermittent hypoxia (AIH) has been demonstrated, through human and animal studies, to be an effective way of increasing spinal motor excitability and strengthening residual synaptic connectivity. AIH utilizes short duration (<2 min) exposures to reduced oxygen levels (~10% inspired oxygen), with alternating exposures to air with normal oxygen levels (~21% inspired oxygen).

Previous publications demonstrate that AIH is a safe and effective intervention to modify motor function in individual with chronic incomplete spinal cord injuries. The use of AIH has been shown to influence the activation in musculature, within 60-120 minutes of administration. In addition, when coupling AIH with overground gait training, an increase in functional endurance, as evaluated through the 6 minute walk test, and gait speed, as evaluated through the 10 meter walk test, were demonstrated. In addition, the use of hypoxic training has been studied in healthy individuals and athletes; however, literature examining the effect of a single bout of AIH on performance is limited.

DETAILED DESCRIPTION:
This study proposes the examine the effects of Acute Intermittent Hypoxia (AIH) in combination with upper extremity training, over the course of a month, to evaluate changes in upper extremity function, dexterity, and ability to complete activities of daily living. The use of acute intermittent hypoxia (AIH) has been demonstrated, through human and animal studies, to be an effective way of increasing spinal motor excitability and strengthening residual synaptic connectivity. AIH utilizes short duration (<2 min) exposures to reduced oxygen levels (~10% inspired oxygen), with alternating exposures to air with normal oxygen levels (~21% inspired oxygen).

Previous publications demonstrate that AIH is a safe and effective intervention to modify motor function in individual with chronic incomplete spinal cord injuries. The use of AIH has been shown to influence the activation in musculature, within 60-120 minutes of administration. In addition, when coupling AIH with overground gait training, an increase in functional endurance, as evaluated through the 6 minute walk test, and gait speed, as evaluated through the 10 meter walk test, were demonstrated. In addition, the use of hypoxic training has been studied in healthy individuals and athletes; however, literature examining the effect of a single bout of AIH on performance is limited.

ELIGIBILITY:
Inclusion Criteria:

* History of a non-progressive spinal cord injury, inclusive of levels of C1-T1.
* Etiology of spinal cord injury is non-progressive in nature
* Be able to demonstrate some hand muscle activation, or use of a tenodesis grasp (wrist extension)
* At least 6 months post injury
* Participants do NOT have to stop taking antispasticity medications to participate in the study.
* Must be tested for anemia with a value of at least 10g/dl (for both men and women).
* Patients will be recommended to their primary care physician to correct anemia if low levels are detected
* Blood pressure must fall within this range- high: 160/110mmHg low: 85/55 mmHg
* Must be asymptomatic (no dizziness, lightheadedness, etc)

Exclusion Criteria:

* Medical conditions, including: congestive heart failure, cardiac arrhythmias, uncontrolled hypertension, uncontrolled diabetes mellitus, chronic obstructive pulmonary disease, emphysema, severe asthma, previous myocardial infraction, or known carotid/intracerebral artery stenosis.
* Women who are currently pregnant or planning on becoming pregnant
* Current tracheostomy placement
* Utilization of mechanical ventilator for breathing
* Current diagnosis of obstructive sleep apnea
* Orthopedic injuries or surgeries that would limit participation
* Concurrent participation in another research study or therapy services
* Comorbid traumatic brain injury or other neurologic injuries that would impact cognition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
GRASSP | 4 weeks
  Graded Redefined Assessment of Strength, Sensation and Prehension

SECONDARY OUTCOMES:
9-hole peg test | 4 weeks
  coordination
grip strength | 4 weeks
  hand strength

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States